CLINICAL TRIAL: NCT03238872
Title: Randomized Controlled Trial of Prompt Mental Health Care
Brief Title: Trial of Prompt Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: The Research Council of Norway (Other); University of Bergen (Other); Göteborg University (Other); Sussex Partnership NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Robert Smith, Researcher, Norwegian Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260659
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Anxiety; Mild to Moderate Depression
Keywords: Anxiety; Depression; CBT; Outcome monitoring; Dissemination; Routine services
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prompt Mental Health Care (Experimental): Clients in the experimental group receive short-term cognitive behavioural therapy in the form of a psycho-educational group course, guided self-help, or individual face-to-face therapy.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Treatment as usual (Active Comparator): Clients in the comparison group are offered treatment as usual from their general practitioner.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy
  Arms: Prompt Mental Health Care
Other: Treatment as usual
  Arms: Treatment as usual

SUMMARY:
Anxiety and depression are among the most common mental disorders in the population. Anxiety and depression have significant consequences at the individual, family and community level, and mental illness is estimated to cost the Norwegian society 180 billion Norwegian kroner annually. The majority of this amount is accounted for by anxiety and depression disorders. Meanwhile, access to mental health services to treat these disorders is limited. The proportion of people who do not receive treatment of those who are in need of treatment is estimated to be over 50%.

Prompt Mental Health Care (PMHC) is a pilot project initiated in 2012 by the Directorate of Health commissioned by the Ministry of Health, with the goal of increasing access to evidence-based treatment for adults with anxiety disorders and mild-to-moderate levels of depression. The treatment offered is cognitive behavioural therapy and should lead to reduced levels of symptoms of anxiety and depression, improved quality of life and better employability. PMHC is based on the English program "Improving Access to Psychological Therapy (IAPT)", which is established in virtually all health communities in England.

The evaluations of IAPT and PMHC have until now been based on relatively weak research designs which make it difficult to know to what extent the initiative really has the desired effect. In this study, PMHC is compared with a control group that receives treatment as usual (often provided by the general practioner) in two PMHC pilot sites (Kristiansand and Sandnes). Participants are randomly assigned to either the PMHC or the control group. The investigators aim to include 1100 clients in the study.

The key objectives of this study are to investigate whether PMHC treatment is more effective as compared to treatment in the control group with regard to symptoms of anxiety and depression, work participation, functional status, and mental well-being. Cost-effectiveness of PMHC is also examined.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9/GAD-7 scores above cut off Level
* Being above 18 years of age and a resident in the pilot sites
* Basic verbal and oral Norwegian proficiency

Exclusion Criteria:

* Entitled to secondary care services due to eating disorder, suicide risk, bipolar disorder, severe depression, invaliding anxiety, psychotic symptoms, severe substance abuse, and personality disorder.
* Two or more previous treatment attempts without effect.
* Serious physical health problem as prime problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Recovery rate | Baseline to 6-month follow-up
  Proportion of clients that have recovered based on predefined cut-offs for the Patient Health Questionnaire (PHQ<10) and Generalized Anxiety Disorder scale (GAD<8).
Changes in mean levels of depression and anxiety | Baseline to 6-month follow-up
  Changes in mean levels of depression and anxiety as measured by respectively PHQ and GAD

SECONDARY OUTCOMES:
Recovery rate / Changes in mean levels of depression and anxiety at 12-month follow-up | Baseline to 12-month follow-up
Recovery rate / Changes in mean levels of depression and anxiety at 24-month and 36-month follow-up, experimental group only. | Baseline to 24/36-month follow-up
Work participation | Baseline to 12-month follow-up
  Increased or maintained work participation at 6 and 12 month follow-up, defined as maintained work participation, new employment or a full or partial return-to-work. Both questionnaire and registry-based data are used for this purpose.
Functional status | Baseline to 12-month follow-up; for experimental group to 36-month follow-up.
  Changes in mean levels of functional status as measured by the Work and Social Adjustment Scale (WSAS).
Health-related quality of life | Baseline to 12-month follow-up; for experimental group to 36-month follow-up.
  Changes in mean levels of health-related quality of life as measured by the EuroQoL-5D (EQ-5D).
Mental Well-being | Baseline to 12-month follow-up; for experimental group to 36-month follow-up.
  Changes in mean levels of mental well-being as measured by the Warwick Edinburgh Mental Well-Being Scale (WEMWBS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smith, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (2):
- Norway (2):
  - Rask Psykisk Helsehjelp Kristiansand, Kristiansand
  - Rask Psykisk Helsehjelp Sandnes, Sandnes

REFERENCES:
- [Derived] Andersen AIO, Knapstad M, Smith ORF. Can registry-based auxiliary variables improve handling of missing outcome data in mental health trials? Evidence from a registry-linked randomized study. Trials. 2025 Dec 9;27(1):33. doi: 10.1186/s13063-025-09346-z. PMID 41366421
- [Derived] Hanevik E, Rovik FMG, Boe T, Knapstad M, Smith ORF. Client predictors of therapy dropout in a primary care setting: a prospective cohort study. BMC Psychiatry. 2023 May 24;23(1):358. doi: 10.1186/s12888-023-04878-7. PMID 37226210
- [Derived] Lervik LV, Hoffart A, Knapstad M, Smith ORF. Exploring the temporal associations between avoidance behavior and cognitions during the course of cognitive behavioral therapy for clients with symptoms of social anxiety disorder. Psychother Res. 2022 Feb;32(2):195-208. doi: 10.1080/10503307.2021.1930243. Epub 2021 Jun 18. PMID 34142636
- [Derived] Knapstad M, Smith ORF. Social anxiety and agoraphobia symptoms effectively treated by Prompt Mental Health Care versus TAU at 6- and 12-month follow-up: Secondary analysis from a randomized controlled trial. Depress Anxiety. 2021 Mar;38(3):351-360. doi: 10.1002/da.23132. Epub 2021 Jan 4. PMID 33393688